CLINICAL TRIAL: NCT03150849
Title: C-X-C Chemokine Receptor 4 as Prognostic Marker in Chronic Lymphocytic Leukemia
Brief Title: C-X-C Chemokine Receptor 4 in Chronic Lymphocytic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed gamal, Principal Investigator, Assiut University
Other Study IDs: cxcll
Record Dates: First submitted 2017-05-07; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient group: patient with chronic lymphocytic leukemia
  Interventions: Diagnostic Test: C-X-C Chemokine Receptor 4
- control group: healthy control group
  Interventions: Diagnostic Test: C-X-C Chemokine Receptor 4

INTERVENTIONS:
Diagnostic Test: C-X-C Chemokine Receptor 4 — marker assessed by flowcytometry in a blood sample

SUMMARY:
Chronic lymphocytic leukemia is the most common type of chronic leukemia, accounting for approximately 40% of all leukemias and mainly affecting older individuals. As it has a highly variable clinical course, identification of molecular and biological prognostic markers has provided new insights into the risk stratification of patients with chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
Prognosis depends primarily on the stage of the disease at diagnosis. There is a correlation between disease stage and median survival. However, about 50% of patients in early stage will develop more advanced disease. Also there is marked variation in disease progression amongst patients with similar Stages .

Extreme clinical heterogeneity is one of the hallmark features of chronic lymphocytic leukemia despite the identification of genetic and phenotypic markers that correlate with prognosis, the biological basis of this clinical variability remains unclear .. In addition, the interactions of chronic lymphocytic leukemia cells with the microenvironment in secondary lymphoid tissues and the bone marrow are known to promote chronic lymphocytic leukemia cell survival and proliferation.

The median age at diagnosis is 72 years, in the last decades chronic lymphocytic leukemia is more often diagnosed also in younger individuals, with almost 15% Of patients Of 55 years old or younger. There is a gender predisposition, As men are more frequently affected by chronic lymphocytic leukemia than women (male: female ratio of 1.5-2:1).

C-X-C chemokine receptor type 4 (CXCR4) is a chemokine and chemokine receptor pair playing critical roles in tumorigenesis. Overexpression of C-X-C chemokine receptor type 4 is a hallmark of many hematological malignancies including acute myeloid leukemia, chronic lymphocytic leukemia and non-Hodgkin's lymphoma, and generally correlates with a poor prognosis. A highly potent competitive antagonist of C-X-C chemokine receptor type 4 recently has been identified with suppression of cancer cells aggressiveness in a variety of cancers.

The protein-coupled receptor C-X-C chemokine receptor type 4 is activated by stromal cell-derived factor 1 and is involved in the control of migration and homing of cells notably for engraftment of normal and neoplastic hematopoietic cells in the bone marrow (BM).

Bruton's tyrosine kinase (BTK) is a key player in B-cell antigen receptor (BCR) signaling that regulates B-cell growth. In addition to B-cell antigen receptor signaling, Bruton's tyrosine kinase participates in signal transduction through growth-factor receptors, Toll-like receptors, integrins and G-protein-coupled receptors such as C-X-C chemokine receptor type 4 and C-X-C chemokine receptor type 5. Bruton's tyrosine kinase inhibition results in impaired C-X-C chemokine receptor type 4 chemokine receptor surface expression, signaling and function in chronic lymphocytic leukemia. inhibition of Bruton's tyrosine kinase function would lead to a loss of tumor volume by preventing replenishment after spontaneous or drug-induced death, and by subverting leukemia cell retention in and homing back to sustaining tissue niches. Decrease C-X-C chemokine receptor type 4 delays disease progression and prolongs survival

ELIGIBILITY:
Inclusion Criteria:

* All patients are newly diagnosed as chronic lymphocytic leukemia

Exclusion Criteria:

* Patients with associated malignancies.
* Chronic lymphocytic leukemia patients on chemotherapy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From Hematology clinic with chronic lynphocytic leukemia
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
The level of C-X-C Chemokine Receptor 4 in chronic lymphocytic leukemia patient and healthy individual | 2 years
  the level of C-X-C Chemokine Receptor 4 marker assessed by flowcytometry in a blood sample

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palmesino E, Moepps B, Gierschik P, Thelen M. Differences in CXCR4-mediated signaling in B cells. Immunobiology. 2006;211(5):377-89. doi: 10.1016/j.imbio.2005.12.003. Epub 2006 Apr 18. PMID 16716807
- [Background] Burger JA, Peled A. CXCR4 antagonists: targeting the microenvironment in leukemia and other cancers. Leukemia. 2009 Jan;23(1):43-52. doi: 10.1038/leu.2008.299. Epub 2008 Nov 6. PMID 18987663
- [Background] Barretina J, Junca J, Llano A, Gutierrez A, Flores A, Blanco J, Clotet B, Este JA. CXCR4 and SDF-1 expression in B-cell chronic lymphocytic leukemia and stage of the disease. Ann Hematol. 2003 Aug;82(8):500-505. doi: 10.1007/s00277-003-0679-0. Epub 2003 May 29. PMID 12783211
- [Background] Marchese A. Endocytic trafficking of chemokine receptors. Curr Opin Cell Biol. 2014 Apr;27:72-7. doi: 10.1016/j.ceb.2013.11.011. Epub 2013 Dec 14. PMID 24680433
- [Background] Domanska UM, Kruizinga RC, Nagengast WB, Timmer-Bosscha H, Huls G, de Vries EG, Walenkamp AM. A review on CXCR4/CXCL12 axis in oncology: no place to hide. Eur J Cancer. 2013 Jan;49(1):219-30. doi: 10.1016/j.ejca.2012.05.005. Epub 2012 Jun 9. PMID 22683307
- [Background] Vlad A, Deglesne PA, Letestu R, Saint-Georges S, Chevallier N, Baran-Marszak F, Varin-Blank N, Ajchenbaum-Cymbalista F, Ledoux D. Down-regulation of CXCR4 and CD62L in chronic lymphocytic leukemia cells is triggered by B-cell receptor ligation and associated with progressive disease. Cancer Res. 2009 Aug 15;69(16):6387-95. doi: 10.1158/0008-5472.CAN-08-4750. Epub 2009 Aug 4. PMID 19654311
- [Background] Li SH, Dong WC, Fan L, Wang GS. Suppression of chronic lymphocytic leukemia progression by CXCR4 inhibitor WZ811. Am J Transl Res. 2016 Sep 15;8(9):3812-3821. eCollection 2016. PMID 27725861